CLINICAL TRIAL: NCT06741215
Title: The Effect of Kinesiophobia on Rehabilitation Outcomes in Patients Undergoing Hand Tendon Surgery
Brief Title: Kinesophobia's Impact on Hand Tendon Rehabilitation
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nadide Koca, Department of Physical Therapy and Rehabilitation, Ankara Training and Research Hospital
Other Study IDs: AnkaraTRH-FTR-NK-01
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Kinesiophobia; Tendon Injuries
Keywords: Tendon Injuries; Kinesiophobia; Hand surgery; Rehabilitation
MeSH Terms: conditions — Kinesiophobia; Tendon Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: High kinesiophobia group: Tampa kinesiophobia score greater than 37
  Interventions: Other: Hand Rehabilitation
- Group 2: Low kinesiophobia group: Tampa kinesiophobia score less than 37
  Interventions: Other: Hand Rehabilitation

INTERVENTIONS:
Other: Hand Rehabilitation — Passive mobilization exercises were initiated for these patients in the first postoperative week.
  Flexor tendon repair patients were immobilized for 3-4 weeks postoperatively. During this period, passive mobilization exercises were with controlled movement. After removing the splint in the third or fourth week, tendon-gliding exercises were initiated, followed by isolated tendon-gliding exercises in the fifth week. Electrotherapy was started in the sixth week (5 days a week, for 15 sessions).
  For extensor tendon repair patients, immobilization lasting 3-6 weeks was applied based on the injury level. During immobilization, passive range of motion (ROM) exercises were performed for adjacent joints while the hand remained in the splint. After splint removal, active and passive ROM exercises, and tendon-gliding exercises with gradually increasing intensity were started according to the injury level. Electrotherapy was started in in the sixth week.

SUMMARY:
Surgically repaired hand tendon injuries may be adversely affected by kinesiophobia during rehabilitation. In this pioneering study, we aimed to investigate the impact of kinesiophobia on functional recovery and rehabilitation outcomes during postoperative rehabilitation of hand tendon injuries.

DETAILED DESCRIPTION:
Patients who underwent primary repair of flexor and/or extensor tendons were included in the study. Data from patients treated with a staged rehabilitation program beginning with passive mobilization in the first week and incorporating electrotherapy and in-person physiotherapy starting from the sixth week were retrospectively analyzed. Patients were grouped as high kinesiophobia (TKS ≥37) or low kinesiophobia (TKS <37) based on their 6th-week assessment. Total Active Motion (TAM) score, Visual Analog Scale (VAS), grip strength, Hand Functional Index (HFI), and Tampa Kinesiophobia Scale (TKS) scores were recorded and statistically compared at the 6th and 12th weeks.

The data of patients who underwent primary tendon repair and received the necessary hand rehabilitation at our hospital were retrospectively analyzed. Passive mobilization exercises were initiated for these patients in the first postoperative week. Flexor tendon repair patients were immobilized for 3-4 weeks postoperatively. During this period, passive mobilization exercises were performed for the metacarpophalangeal (MCP), proximal interphalangeal (PIP), and distal interphalangeal (DIP) joints with controlled movement. After removing the splint in the third or fourth week, tendon-gliding exercises were initiated, followed by isolated tendon-gliding exercises in the fifth week. Electrotherapy was started in the sixth week (5 days a week, for 15 sessions), including hydromassage, pulsed ultrasound, transcutaneous electrical nerve stimulation (TENS), and hot pack therapy. Gentle stretching exercises were performed on joints with ROM limitations. Light resistance exercises were introduced during the 7th-8th week, and strengthening exercises with daily-use weights were started in the 10th-12th week.

For extensor tendon repair patients, immobilization lasting 3-6 weeks was applied based on the injury level. During immobilization, passive range of motion (ROM) exercises were performed for adjacent joints while the hand remained in the splint. After splint removal, active and passive ROM exercises, and tendon-gliding exercises with gradually increasing intensity were started according to the injury level. Electrotherapy and in-person physiotherapy began in the sixth week, and gentle stretching for joints with ROM limitations and strengthening exercises were introduced starting in the 8th-10th week.

The data included the patient's age, sex, occupation, type of injury, injury level, time elapsed since the injury, dominant hand, duration of splint use, and the treatment methods applied. Additionally, at the 6th and 12th weeks, pre- and post-physiotherapy measurements of range of motion (ROM), Visual Analog Scale (VAS) scores, Hand Functional Index (HFI) scores, Tampa Kinesiophobia Scale (TKS) scores, and hand grip (HG) strength scores were recorded.

Finger ROM measurements were performed using a finger goniometer. ROM values for the affected finger's MCP, PIP, and DIP joints were recorded. The measured ROM values were evaluated according to the Total Active Motion (TAM) scoring system of the American Society for Surgery of the Hand. TAM is calculated by subtracting the total extension lag from the sum of active flexion angles of the affected finger's MCP, PIP, and DIP joints. Each patient's pre- and post-treatment TAM values were calculated and recorded [Collocott SJF, Kelly E, Foster M, Myhr H, Wang A, Ellis RF. A randomized clinical trial comparing early active motion programs: Earlier hand function, TAM, and orthotic satisfaction with a relative motion extension program for zones V and VI extensor tendon repairs. J Hand Ther. 2020;33(1):13-24.].

Pain severity was assessed pre- and post-treatment using the VAS. In this scale, where 0 indicates no pain, and 10 indicates the most severe pain, patients were asked to rate their pain on a line from 0 to 10. VAS is a simple, valid, and reliable method commonly used to assess pain in studies. Pain severity was categorized as follows: VAS 1-4 (mild pain), VAS 5-6 (moderate pain), and VAS 7-10 (severe pain) [Bodian CA, Freedman G, Hossain S, Eisenkraft JB, Beilin Y. The visual analog scale for pain: clinical significance in postoperative patients. Anesthesiology. 2001 Dec;95(6):1356-61.].

The HFI consists of 9 questions evaluating wrist and finger movements. The first question is scored from 0-3 (0=performs the movement completely with normal speed, 1=delayed performance, 2=partial performance, 3=unable to perform), while questions 2, 3, 4, 5, 8, and 9 are scored from 0-2 (0=performs the movement completely, 1=performs with difficulty and delay, 2=unable to perform). Questions 6 and 7 are scored from 1-3 (1=performs the movement completely, 2=performs with difficulty and delay, 3=partial performance). The total score ranges from 2 to 21, with higher scores indicating worse hand function [Lefevre-Colau MM, Poiraudeau S, Fermanian J, Etchepare F, Alnot JY, Le Viet D, Leclercq C, Oberlin C, Bargy F, Revel M. Responsiveness of the Cochin rheumatoid hand disability scale after surgery. Rheumatology (Oxford). 2001;40(8):843-50.].

Kinesiophobia was assessed using the Turkish version of the TSK. This scale consists of 17 items measuring fear of movement and/or reinjury. It evaluates fear-avoidance parameters in daily activities with statements such as, "I am afraid of injuring myself if I exercise," "I cannot do what normal people do because I injure myself too easily," and "My body will always be at risk because of what happened to me." Patients respond to these statements by selecting one of the options: strongly disagree, disagree, agree, or strongly agree, scored as 1-4, respectively. Items 4, 8, 12, and 16 are reverse scored, and the total score ranges from 17 to 68, with higher scores indicating higher levels of kinesiophobia. A threshold score of 37 was used to classify patients: those with Tampa scores ≥37 were categorized as the high-kinesiophobia group. In contrast, those with scores <37 were categorized as the low-kinesiophobia group [Tuna Z, Oskay D. Fear of movement and its effects on hand function after tendon repair. Hand Surg Rehabil. 2018:S2468-1229(18)30092-6.].

ELIGIBILITY:
Inclusion Criteria:

• Clinical diagnosis of underwent primary repair for flexor and/or extensor tendon injuries

Exclusion Criteria:

* Patients with associated fractures
* Peripheral nerve and vascular injuries
* Rheumatoid arthritis
* Diabetes mellitus
* Peripheral artery disease
* Other rheumatic diseases affecting the hand

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent primary repair of flexor and/or extensor tendon injuries
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Tampa Scale of Kinesiophobia (TSK) scores | six week
  The original Tampa Scale of Kinesiophobia (TKS) was developed by Miller, Kopri and Todd in 1991 but was not published [Miller R., Kori S., Todd D. The Tampa Scale: a measure of kinesiophobia. Clin J Pain. 1991;7(1):51-52.]. TKS is a 17-item scale developed to measure fear of movement/reinjury. The scale includes parameters of injury/reinjury and fear-avoidance in work-related activities. We used the Turkish version in our study. [Acar S., Savci S., Keskinoğlu P., Akdeniz B., Özpelit E., Özcan Kahraman B., Karadibak D., Sevinc C. Tampa Scale of Kinesiophobia for Heart Turkish Version Study: cross-cultural adaptation, exploratory factor analysis, and reliability. J Pain Res. 2016 Jun 23;9:445-51.]

SECONDARY OUTCOMES:
Visual analog scale (VAS) scores | six week
  Pain severity was assessed pre- and post-treatment using the VAS. In this scale, where 0 indicates no pain, and 10 indicates the most severe pain, patients were asked to rate their pain on a line from 0 to 10. VAS is a simple, valid, and reliable method commonly used to assess pain in studies. Pain severity was categorized as follows: VAS 1-4 (mild pain), VAS 5-6 (moderate pain), and VAS 7-10 (severe pain). [Bodian CA, Freedman G, Hossain S, Eisenkraft JB, Beilin Y. The visual analog scale for pain: clinical significance in postoperative patients. Anesthesiology. 2001 Dec;95(6):1356-61.]
Total Active Motion (TAM) | six week
  TAM is calculated by subtracting the total extension lag from the sum of active flexion angles of the affected finger's MCP, PIP, and DIP joints. Each patient's pre- and post-treatment TAM values were calculated and recorded [Collocott SJF, Kelly E, Foster M, Myhr H, Wang A, Ellis RF. A randomized clinical trial comparing early active motion programs: Earlier hand function, TAM, and orthotic satisfaction with a relative motion extension program for zones V and VI extensor tendon repairs. J Hand Ther. 2020;33(1):13-24.]
Hand Functional Index (HFI) scores | six week
  The HFI consists of 9 questions evaluating wrist and finger movements. The first question is scored from 0-3 (0=performs the movement completely with normal speed, 1=delayed performance, 2=partial performance, 3=unable to perform), while questions 2, 3, 4, 5, 8, and 9 are scored from 0-2 (0=performs the movement completely, 1=performs with difficulty and delay, 2=unable to perform). Questions 6 and 7 are scored from 1-3 (1=performs the movement completely, 2=performs with difficulty and delay, 3=partial performance). The total score ranges from 2 to 21, with higher scores indicating worse hand function [Lefevre-Colau MM, Poiraudeau S, Fermanian J, Etchepare F, Alnot JY, Le Viet D, Leclercq C, Oberlin C, Bargy F, Revel M. Responsiveness of the Cochin rheumatoid hand disability scale after surgery. Rheumatology (Oxford). 2001;40(8):843-50.].

CONTACTS AND LOCATIONS:
Overall Officials: Nadide Koca, M.D., Principal Investigator — Department of Physical Therapy and Rehabilitation, University of Health Sciences
Locations (1):
- Department of Physical Therapy and Rehabilitation, University of Health Sciences, Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collocott SJF, Kelly E, Foster M, Myhr H, Wang A, Ellis RF. A randomized clinical trial comparing early active motion programs: Earlier hand function, TAM, and orthotic satisfaction with a relative motion extension program for zones V and VI extensor tendon repairs. J Hand Ther. 2020 Jan-Mar;33(1):13-24. doi: 10.1016/j.jht.2018.10.003. Epub 2019 Mar 21. PMID 30905495
- [Background] Cai L, Liu Y, Xu H, Xu Q, Wang Y, Lyu P. Incidence and Risk Factors of Kinesiophobia After Total Knee Arthroplasty in Zhengzhou, China: A Cross-Sectional Study. J Arthroplasty. 2018 Sep;33(9):2858-2862. doi: 10.1016/j.arth.2018.04.028. Epub 2018 Apr 23. PMID 29776855
- [Background] Bodian CA, Freedman G, Hossain S, Eisenkraft JB, Beilin Y. The visual analog scale for pain: clinical significance in postoperative patients. Anesthesiology. 2001 Dec;95(6):1356-61. doi: 10.1097/00000542-200112000-00013. PMID 11748392
- [Background] Bordeleau M, Vincenot M, Lefevre S, Duport A, Seggio L, Breton T, Lelard T, Serra E, Roussel N, Neves JFD, Leonard G. Treatments for kinesiophobia in people with chronic pain: A scoping review. Front Behav Neurosci. 2022 Sep 20;16:933483. doi: 10.3389/fnbeh.2022.933483. eCollection 2022. PMID 36204486
- [Background] Bilgin S, Cetin H, Karakaya J, Kose N. Multivariate Analysis of Risk Factors Predisposing to Kinesiophobia in Persons With Chronic Low Back and Neck Pain. J Manipulative Physiol Ther. 2019 Oct;42(8):565-571. doi: 10.1016/j.jmpt.2019.02.009. Epub 2019 Nov 23. PMID 31771838
- [Background] Bennett DJ, Bango J, Rothkopf DM. Hand Therapy after Flexor and Extensor Tendon Repair: Assessing Predictors of Loss to Follow-up. Plast Reconstr Surg Glob Open. 2023 Apr 26;11(4):e4941. doi: 10.1097/GOX.0000000000004941. eCollection 2023 Apr. PMID 37124389
- [Background] Bartlett O, Farnsworth JL. The Influence of Kinesiophobia on Perceived Disability in Patients With an Upper-Extremity Injury: A Critically Appraised Topic. J Sport Rehabil. 2021 Mar 3;30(5):818-823. doi: 10.1123/jsr.2020-0179. PMID 33662934
- [Background] Alshahrani MS, Reddy RS. Kinesiophobia, limits of stability, and functional balance assessment in geriatric patients with chronic low back pain and osteoporosis: a comprehensive study. Front Neurol. 2024 Feb 13;15:1354444. doi: 10.3389/fneur.2024.1354444. eCollection 2024. PMID 38414551
- [Background] Alshahrani MS, Reddy RS, Tedla JS, Asiri F, Alshahrani A. Association between Kinesiophobia and Knee Pain Intensity, Joint Position Sense, and Functional Performance in Individuals with Bilateral Knee Osteoarthritis. Healthcare (Basel). 2022 Jan 7;10(1):120. doi: 10.3390/healthcare10010120. PMID 35052284
- [Background] Alito A, Cifalino ME, Fontana JM, Verme F, Pitera P, Capodaglio P. Tackling Kinesiophobia in Chronic Shoulder Pain: A Case Report on the Combined Effect of Pain Education and Whole-Body Cryostimulation. J Clin Med. 2024 Apr 3;13(7):2094. doi: 10.3390/jcm13072094. PMID 38610859
- [Background] Aleksic M, Selakovic I, Tomanovic Vujadinovic S, Kadija M, Milovanovic D, Meissner W, Zaslansky R, Sreckovic S, Dubljanin-Raspopovic E. Understanding Kinesiophobia: Predictors and Influence on Early Functional Outcomes in Patients with Total Knee Arthroplasty. Geriatrics (Basel). 2024 Aug 13;9(4):103. doi: 10.3390/geriatrics9040103. PMID 39195133
- [Background] Al-Amiry B, Rahim A, Knutsson B, Mattisson L, Sayed-Noor A. Kinesiophobia and its association with functional outcome and quality of life 6-8 years after total hip arthroplasty. Acta Orthop Traumatol Turc. 2022 Jul;56(4):252-255. doi: 10.5152/j.aott.2022.21318. PMID 35968616
- [Background] Lefevre-Colau MM, Poiraudeau S, Fermanian J, Etchepare F, Alnot JY, Le Viet D, Leclercq C, Oberlin C, Bargy F, Revel M. Responsiveness of the Cochin rheumatoid hand disability scale after surgery. Rheumatology (Oxford). 2001 Aug;40(8):843-50. doi: 10.1093/rheumatology/40.8.843. PMID 11511751
- [Background] Duruoz MT, Cerrahoglu L, Dincer-Turhan Y, Kursat S. Hand function assessment in patients receiving haemodialysis. Swiss Med Wkly. 2003 Aug 9;133(31-32):433-8. doi: 10.4414/smw.2003.10216. PMID 14562186
- [Background] Osteras N, Risberg MA, Kvien TK, Engebretsen L, Nordsletten L, Bruusgaard D, Schjervheim UB, Haugen IK, Hammer HB, Provan S, Oiestad BE, Semb AG, Rollefstad S, Hagen KB, Uhlig T, Slatkowsky-Christensen B, Kjeken I, Flugsrud G, Grotle M, Sesseng S, Edvardsen H, Natvig B. Hand, hip and knee osteoarthritis in a Norwegian population-based study--the MUST protocol. BMC Musculoskelet Disord. 2013 Jul 5;14:201. doi: 10.1186/1471-2474-14-201. PMID 23826721
- [Background] Guney-Deniz H, Irem Kinikli G, Caglar O, Atilla B, Yuksel I. Does kinesiophobia affect the early functional outcomes following total knee arthroplasty? Physiother Theory Pract. 2017 Jun;33(6):448-453. doi: 10.1080/09593985.2017.1318988. Epub 2017 May 8. PMID 28481125
- [Background] Filardo G, Merli G, Roffi A, Marcacci T, Berti Ceroni F, Raboni D, Bortolotti B, Kon E, Marcacci M. Kinesiophobia and depression affect total knee arthroplasty outcome in a multivariate analysis of psychological and physical factors on 200 patients. Knee Surg Sports Traumatol Arthrosc. 2017 Nov;25(11):3417-3423. doi: 10.1007/s00167-016-4201-3. Epub 2016 Jun 21. PMID 27329175
- [Background] Tuna Z, Oskay D, Gokkurt A, Mete O, Baglan Yentur S, Ambarcioglu P. Does earlier splint removal truly affect functional recovery and kinesiophobia after tendon repair? Hand Surg Rehabil. 2020 Sep;39(4):310-315. doi: 10.1016/j.hansur.2020.01.006. Epub 2020 Feb 20. PMID 32088423
- [Background] Das De S, Vranceanu AM, Ring DC. Contribution of kinesophobia and catastrophic thinking to upper-extremity-specific disability. J Bone Joint Surg Am. 2013 Jan 2;95(1):76-81. doi: 10.2106/JBJS.L.00064. PMID 23283376